CLINICAL TRIAL: NCT05985382
Title: Comparing the Effects of Upper and Lower Body Resistance Training on Pain Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Abigail Wilson, Assistant Professor, University of Central Florida
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower Body Resistance Exercise (Experimental): Participants will perform a leg extension exercise with weight that is 75% of their estimated 1-repetition maximum (1-RM) for 3 sets of 10 repetitions.
  Interventions: Other: Lower Body Resistance Exercise
- Upper Body Resistance Exercise (Experimental): Participants will perform a shoulder press with weight that is 75% of their estimated 1-repetition maximum (1-RM) for 3 sets of 10 repetitions.
  Interventions: Other: Upper Body Resistance Exercise

INTERVENTIONS:
Other: Lower Body Resistance Exercise — Participants will complete a leg extension exercise with weight equivalent to 75% of their estimated 1-repetition maximum 3 sets, 10 repetitions.
  Arms: Lower Body Resistance Exercise
Other: Upper Body Resistance Exercise — Participants will complete a leg extension exercise with weight equivalent to 75% of their estimated 1-repetition maximum 3 sets, 10 repetitions.
  Arms: Upper Body Resistance Exercise

SUMMARY:
Resistance exercise may immediately lessen the perception of pain. The purpose of this study is compare the effects of an upper body exercise to a lower body exercise on the perception of pain (pressure pain threshold).

ELIGIBILITY:
Inclusion Criteria:

* pain free

Exclusion Criteria:

* non-English speaking
* regular use of prescription pain medications
* current or history of chronic pain condition
* currently taking blood-thinning medication
* any blood clotting disorder
* medical conditions known to affect sensation, such as: uncontrolled diabetes or neurological conditions
* any contraindication to the application of ice, including: uncontrolled hypertension, cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, circulatory compromise
* not physically ready to exercise without a medical exam as indicated by the Physical Activity Readiness Questionnaire Plus (PAR-Q+)
* surgery, injury, or fracture within the past 6 months
* unable to perform exercise portions of the study
* unable to attend three sessions
* pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Wilson, PT, DPT, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Lower Then Upper Body Resistance Exercise: Participants will perform a lower body resistance exercise first then upper body resistance exercise. This is a cross-over design.
  Lower Body Resistance Exercise: Participants will complete a leg extension exercise with weight equivalent to 75% of their estimated 1-repetition maximum 3 sets, 10 repetitions.
  Participants will perform a shoulder press with weight that is 75% of their estimated 1-repetition maximum (1-RM) for 3 sets of 10 repetitions.
  Upper Body Resistance Exercise: Participants will complete a leg extension exercise with weight equivalent to 75% of their estimated 1-repetition maximum 3 sets, 10 repetitions.
- Upper Then Lower Body Resistance Exercise: Participants will perform a upper body resistance exercise first then upper body resistance exercise. This is a cross-over design.
  Upper Body Resistance Exercise: Participants will complete a leg extension exercise with weight equivalent to 75% of their estimated 1-repetition maximum 3 sets, 10 repetitions.
  Lower Body Resistance Exercise: Participants will complete a leg extension exercise with weight equivalent to 75% of their estimated 1-repetition maximum 3 sets, 10 repetitions.
  Participants will perform a shoulder press with weight that is 75% of their estimated 1-repetition maximum (1-RM) for 3 sets of 10 repetitions.
Period: Overall Study
Arm/Group | Lower Then Upper Body Resistance Exercise | Upper Then Lower Body Resistance Exercise
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- Upper and Lower Body Resistance Exercise: All participants will perform a leg extension exercise with weight that is 75% of their estimated 1-repetition maximum (1-RM) for 3 sets of 10 repetitions.
  Lower Body Resistance Exercise: Participants will complete a leg extension exercise with weight equivalent to 75% of their estimated 1-repetition maximum 3 sets, 10 repetitions.
  Participants will perform a shoulder press with weight that is 75% of their estimated 1-repetition maximum (1-RM) for 3 sets of 10 repetitions.
  Upper Body Resistance Exercise: Participants will complete a leg extension exercise with weight equivalent to 75% of their estimated 1-repetition maximum 3 sets, 10 repetitions.
Arm/Group | Upper and Lower Body Resistance Exercise
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Lower Body Resistance Exercise
Description: For pressure pain threshold, an algometer was gradually increased until the sensation changed from pressure to pain. Pressure at threshold was recorded in kilopascals.
Time Frame: Pressure pain threshold will be applied to the quadriceps immediately after each exercise.
Measure: Mean (Standard Deviation); unit: kilopascals
Arm/Group | Lower Body Resistance Exercise | Upper Body Resistance Exercise
Number analyzed (Participants) | 30 | 30
kilopascals | 594.10 (234.74) | 572.54 (249.87)

2. Secondary Outcome: Heat Pain Threshold
Description: All participants completed Heat Pain Threshold. For heat pain threshold, a thermode will gradually warm up from 32 degrees Celsius until the participant reports the sensation changes from comfortable warmth to slightly unpleasant pain. The temperature at threshold will be recorded.
Time Frame: Heat Pain Threshold will be applied over the quadriceps before and after the exercise.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Lower Body Resistance Exercise | Upper Body Resistance Exercise
Number analyzed (Participants) | 30 | 30
Degrees Celsius | 43.75 (3.27) | 43.56 (3.18)

ADVERSE EVENTS:
Time Frame: Adverse events were not collected.
Description: Adverse events were not collected
Groups:
- Lower Body Then Upper Body Resistance Exercise: Participants will perform a leg extension exercise with weight that is 75% of their estimated 1-repetition maximum (1-RM) for 3 sets of 10 repetitions.
  Lower Body Resistance Exercise: Participants will complete a leg extension exercise with weight equivalent to 75% of their estimated 1-repetition maximum 3 sets, 10 repetitions.
- Upper Body Then Lower Body Resistance Exercise: Participants will perform a shoulder press with weight that is 75% of their estimated 1-repetition maximum (1-RM) for 3 sets of 10 repetitions.
  Upper Body Resistance Exercise: Participants will complete a leg extension exercise with weight equivalent to 75% of their estimated 1-repetition maximum 3 sets, 10 repetitions.
Arm/Group | Lower Body Then Upper Body Resistance Exercise | Upper Body Then Lower Body Resistance Exercise
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT05985382/Prot_SAP_000.pdf